CLINICAL TRIAL: NCT01228006
Title: Study for Effectiveness Evaluation of Panax Ginseng, Vitamins and Minerals (Natugerin®) in Improvement of Stress and Fatigue
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NATEMS0310; Version 02 - March 11, 2010
Record Dates: First submitted 2010-04-08; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Stress; Fatigue
Keywords: Reduction of stress and fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): NatusGerin
  Interventions: Dietary Supplement: NatusGerin
- Control (Placebo Comparator): Gelatin capsules identical to drug test
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Dietary Supplement: NatusGerin — 1 capsule, 2 times a day.
  Arms: Treatment
Other: Placebo capsules — 1 capsule, 2 times a day
  Arms: Control

SUMMARY:
It is hoped that the group treated with Panax Ginseng, Vitamins and Minerals obtain significant reduction in levels of stress and fatigue and that the results are superior to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Agree with all study procedures, signing the IC in two ways, by his own free will;
* Patients older than 18 years, male or female, regardless of ethnicity or social class;
* Presence of pictures of mild to moderate stress, confirmed with the aid of the Stress Symptom Inventory (ISS), which considers stress and mild to moderate classification Alert classification Resistance;
* Presence frame of fatigue with a score greater than 36 according to the Fatigue Severity Scale (FSS).

Exclusion Criteria:

* Participation in clinical trials in the 12 months preceding the survey;
* Current treatment with drugs that are stimulants or central nervous system depressants such as hypnotics, anxiolytics, antipsychotics, antidepressants, statins and muscle relaxants;
* Alternative Therapies that scientifically, or have no influence in the tables of stress or fatigue as acupuncture or relaxing massages;
* Treatment psychotherapeutic medication or not;
* Current treatment or prediction of treatment with oral anticoagulants (due to interaction with the tocopherol);
* Women who are pregnant or lactating;
* Patients with lactose intolerance;
* Patients allergic to soy or peanuts;
* chronic renal failure;
* Patients using other multivitamins or individual vitamins such as vitamin D and / or A.
* Chronic alcoholism;
* Patients with clinical diagnosis of diseases causing severe chronic pain or adversely affect the clinical interpretation as fibromyalgia, multiple sclerosis, neuropathies and myopathies;
* Patients with hypothyroidism or hyperthyreosis diagnosed clinically;
* Patient history and physical examination suggestive of severe hepatorenal failure;
* Patients with decompensated diabetes mellitus (fasting glucose above 180 mg / dL);
* Patients being treated for cancer;
* Amendment of the routine of life during the study as early vacation or suspected change in working hours;
* Patients with complaints of excessive sleepiness caused by organic source frameworks such as sleep apnea and morbid obesity (BMI above 35);
* History of hypersensitivity to any component of the product under investigation;
* Any finding of clinical observation (clinical history or physical examination) that is interpreted by the physician investigator as a risk to the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of the product Natus Gerin, compared to placebo, ® in improving symptoms of stress and fatigue in patients with clinical diagnosis of mild to moderate stress | 14 and 28 days

SECONDARY OUTCOMES:
Improvement in quality of sexual function. | 14 and 28 days
Improvement in quality of life. | 14 and 28 days.
Decrease stress during treatment (28 days) | 14 and 28 days
Decrease fatigue during treatment (28 days) | 14 and 28 days